CLINICAL TRIAL: NCT06249386
Title: Adapting and Piloting Behavioral Activation for Veterans With Co-Occurring AUD and Posttraumatic Stress Disorder
Brief Title: Adapting and Piloting Behavioral Activation for Veterans With Alcohol Use Disorder and Posttraumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Duke University (Other)
Responsible Party: Principal Investigator, Shannon Blakey, Research Clinical Psychologist, RTI International
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0219135; R34AA030820 (NIH); Pro00113641 (Other: Duke University School of Medicine); STUDY00022679 (Other: RTI International)
Record Dates: First submitted 2024-01-30; First posted 2024-02-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder; Posttraumatic Stress Disorder
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic | interventions — Secondary Prevention

STUDY DESIGN:
Intervention Model Description: Participants will be block randomized to either Behavioral Activation treatment (n=23) or Relapse Prevention treatment (n=23).
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blind to treatment condition. The participant, study therapist, and PI (providing clinical consultation and evaluating therapist fidelity to treatment protocol) will not be blinded to participants' assigned treatment condition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Activation (BA) (Experimental): Individual psychotherapy
  Interventions: Behavioral: Behavioral Activation (BA)
- Relapse Prevention (RP) (Active Comparator): Individual psychotherapy
  Interventions: Behavioral: Relapse Prevention (RP)

INTERVENTIONS:
Behavioral: Behavioral Activation (BA) — BA reduces alcohol use and posttraumatic stress symptoms and increases psychosocial functioning via psychoeducation, activity monitoring, values clarification, and activity scheduling.
  Arms: Behavioral Activation (BA)
Behavioral: Relapse Prevention (RP) — RP reduces alcohol use via increasing awareness and avoidance of high-risk situations, enhancing drink refusal skills, improving assertiveness, and other strategies.
  Arms: Relapse Prevention (RP)

SUMMARY:
The goal of this clinical trial is to compare an adaptation of Behavioral Activation, a behavioral intervention, to Relapse Prevention treatment, another behavioral intervention, in a sample of U.S. military veterans with co-occurring alcohol use disorder (AUD) and posttraumatic stress disorder (PTSD).

The primary aims of this study are to:

1. Adapt Behavioral Activation to treat veterans with AUD/PTSD,
2. Evaluate the feasibility, acceptability, and preliminary effects of Behavioral Activation for AUD/PTSD, and
3. Explore geospatial analysis as a new method for measuring AUD/PTSD recovery.

Participants will complete self-report and interview measures immediately before and immediately after treatment. Participants will also be asked to participate in passive geospatial assessment for 14-day periods immediately before and immediately after treatment. Participants will be randomized to treatment condition, which involves 8 sessions of either Behavioral Activation or Relapse Prevention, delivered individually by a trained study therapist.

DETAILED DESCRIPTION:
Alcohol use disorder (AUD) frequently co-occurs with posttraumatic stress disorder (PTSD) among U.S. military veterans. Compared to veterans with AUD only, veterans with AUD/PTSD have greater symptom severity, more psychosocial functioning difficulties, and higher risk of suicide. Many people with AUD/PTSD perform behaviors aimed at avoiding unpleasant emotions (e.g., drinking to avoid trauma-related nightmares, skipping social events to avoid anxiety-provoking crowds). These "avoidance behaviors" provide temporary relief from unpleasant emotions, but they maintain AUD/PTSD and interfere with long-term functioning. Although treatments for AUD/PTSD exist, they emphasize symptom reduction (not functional improvement) and have dropout rates as high as 50%. Originally developed to treat depression, Behavioral Activation (BA) is an intervention that increases daily participation in rewarding, alcohol-free activities relevant to patients' social, vocational, and health-related values. Randomized controlled trials (RCTs) adapting BA for other disorders have shown that BA is efficacious for adults with alcohol/drug use disorders and acceptable to veterans with PTSD, but BA has not been used to treat co-occurring AUD/PTSD. Additionally, because RCTs of AUD/PTSD treatments typically emphasize significant mean group differences in AUD/PTSD outcomes, less is known about the degree to which these treatments yield clinically significant improvements at the individual level. Individual-level improvements in AUD/PTSD should be evident not only in subjective clinical assessments, but also in objective measures of geospatial activity. Specifically, patients' daily geospatial activity is likely to change as they decrease their avoidance behaviors and increase their engagement in various social, vocational, and health-promoting activities. Advances in geospatial methods, coupled with discreet and portable global positioning system (GPS) trackers, have made it possible to objectively measure people's spatial movement within their communities. Yet although geospatial methods have been used to identify social determinants of alcohol use, they have not been used to measure response to AUD or AUD/PTSD treatment. As the long-term objectives of this work are to identify a more acceptable AUD/PTSD treatment option and improve the measurement of AUD/PTSD recovery, this R34 project will address the following specific aims: (1) adapt BA for use with veterans with AUD/PTSD; (2) evaluate the feasibility, acceptability, and preliminary effects of BA, relative to Relapse Prevention, for veterans with AUD/PTSD in a pilot RCT; and (3) explore geospatial analysis of GPS-collected data as a new approach to measuring AUD/PTSD treatment response. This study will advance research and practice by piloting a novel application of BA and a novel measure of AUD/PTSD recovery. This project aligns with the National Institute on Alcohol Abuse and Alcoholism's special interest in investigating treatments for patients with AUD and co-occurring disorders, dimensions of functioning and well-being associated with recovery, and innovative methods for evaluating AUD treatment and recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Be a U.S. veteran,
2. Be at least 18 years old,
3. Meet Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for current AUD,
4. Report 3+ heavy drinking days (5+ drinks for men/4+ drinks for women) or 1+ heavy drinking week (15+ drinks men/8+ drinks women) in the past 30 days,
5. Meet DSM-5 criteria for current PTSD or satisfy the definition of current subthreshold PTSD (i.e., up to one of symptom clusters B-E may fall below diagnostic threshold),
6. Be fluent and literate in English, and
7. Be able to provide voluntary, informed consent to participate.

Exclusion Criteria:

1. Current mania/hypomania or current psychosis,
2. Lifetime alcohol withdrawal-related seizures, delirium, or hallucinations,
3. Prior inpatient alcohol withdrawal management,
4. Current DSM-5 severe drug use disorder (DUD) except for severe tobacco use disorder,
5. Psychotropic (including alcohol abstinence) medication changes within 30 days of study enrollment or plans to change medications during the study,
6. Current/planned non-study BA for any disorder during the study, or
7. Current/planned evidence-based psychotherapy for AUD, PTSD, or DUD during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-01-17 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
Timeline Follow-Back (alcohol use) | Through study completion, an average of 3 months
  Changes in past-30-day alcohol consumption from baseline to immediately post-treatment
Clinician-Administered PTSD Scale for DSM-5 (PTSD severity) | Through study completion, an average of 3 months
  Changes in past-month PTSD severity from baseline to immediately post-treatment

SECONDARY OUTCOMES:
Brief Inventory of Psychosocial Functioning (psychosocial functioning) | Through study completion, an average of 3 months
  Changes in past-30-day psychosocial functioning from baseline to immediately post-treatment
Geospatial activity | Through study completion, an average of 3 months
  Changes in past-14-day geospatial activity metrics (e.g., activity space) from baseline to immediately post-treatment
PTSD Checklist for DSM-5 (PCL-5) | Through study completion, an average of 3 months
  Changes in past-month PTSD severity from baseline to immediately post-treatment
Generalized Anxiety Disorder-7 (GAD-7) | Through study completion, an average of 3 months
  Changes in past-2-week anxiety severity from baseline to immediately post-treatment
Patient Health Questionnaire-9 (PHQ-9) | Through study completion, an average of 3 months
  Changes in past-2-week depressive symptom severity from baseline to immediately posttreatment
Insomnia Severity Index | Through study completion, an average of 3 months
  Changes in past-2-week sleep disturbance from baseline to immediately post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shannon M Blakey, PhD, Principal Investigator — RTI International; Eric B Elbogen, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University School of Medicine, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from consenting participants will be submitted to the National Institute on Alcohol Abuse and Alcoholism Data Archive.
Time Frame: All collection data are shared automatically two years after the grant end date specified on the first Notice of Award. PI requests for exceptions will be considered for only extreme and unusual circumstances (e.g., unanticipated life event [death of family member] or other force majeure).
Access Criteria: Data access requires sponsorship by an Institution on behalf of Recipient(s) and satisfaction of any other criteria required by the National Institute on Alcohol Abuse and Alcoholism Data Archive.

REFERENCES:
- [Derived] Blakey SM, Alsobrooks AK, Morgan-Lopez AA, Kruskamp N, Simpson TL, Daughters SB, DuBois CM, Huang JS, Evans J, Serrano BN, Calhoun PS, Beckham JC, Elbogen EB. Behavioral activation for veterans with co-occurring alcohol use disorder and posttraumatic stress disorder: Basis and methodology for a pilot randomized controlled trial. Contemp Clin Trials. 2024 Nov;146:107670. doi: 10.1016/j.cct.2024.107670. Epub 2024 Aug 24. PMID 39186971